CLINICAL TRIAL: NCT00860275
Title: A Study of the Effect of Concomitant Administration of Ketoconazole or Fluconazole on the Pharmacokinetics of BMS-708163 in Healthy Subjects
Brief Title: Drug-Drug Interaction (DDI) w/Ketoconazole or Fluconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CN156-019
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2009-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BMS 708163; Ketoconazole; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMS-708163 / Ketoconazole (Active Comparator)
  Interventions: Drug: BMS-708163; Drug: BMS-708163 + Ketoconazole; Drug: Ketoconazole
- BMS-708163 / Fluconazole (Active Comparator)
  Interventions: Drug: BMS-708163; Drug: Fluconazole; Drug: BMS-708163 + Fluconazole

INTERVENTIONS:
Drug: BMS-708163 — Capsule, Oral, 50 mg, once, Day 1
Drug: BMS-708163 + Ketoconazole — (BMS-708163) - Capsule, Oral, 50 mg, daily, 1 day Day 12 (Ketoconazole) - Tablet, Oral, 400 mg, daily, 1 day
  Arms: BMS-708163 / Ketoconazole
Drug: Ketoconazole — Tablet, Oral, 400 mg, daily, 16 days
  Arms: BMS-708163 / Ketoconazole
Drug: Fluconazole — Tablet, Oral, 1 day 400 mg then 3 days 200 mg
  Arms: BMS-708163 / Fluconazole
Drug: BMS-708163 + Fluconazole — (BMS-708163) - Capsule, Oral, 50 mg, daily, 1 day (Day 12) (Fluconazole) - Tablet, Oral, 200 mg, daily, 13 days
  Arms: BMS-708163 / Fluconazole

SUMMARY:
The purpose of the study is to determine if the concomitant administration of either ketoconazole or fluconazole with BMS-708163 will affect the PK of BMS-708163 and to assess safety and tolerability of BMS-708163

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and postmenopausal female subjects 18-55 yrs old inclusive

Exclusion:

* Premenopausal women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
PK profile of BMS-708163 | Within 14 days after dose

SECONDARY OUTCOMES:
Safety and tolerability of BMS-708163 when administered alone and with either ketoconazole or fluconazole | During the entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx